CLINICAL TRIAL: NCT02975570
Title: Prospective, Randomized, Open Label Phase 3 Study of the Efficacy and Tolerability of Delamanid, Linezolid, Pyrazinamide and Levofloxacin for Treatment of Patients With Fluoroquinolone-susceptible Multidrugresistant--Tuberculosis (MDR-TB)
Brief Title: Efficacy and Tolerability of Delamanid, Linezolid, Pyrazinamide and Levofloxacin
Acronym: DAZZLE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study could not be conducted since funding was not obtained.
Sponsor: Boston University (Other)
Collaborators: Westat (Other); University of Florida (Other)
Responsible Party: Principal Investigator, Charles R Horsburgh, Professor of Epidemiology, Boston University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-36160
Record Dates: First submitted 2016-10-21; First posted 2016-11-29 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Tuberculosis Multi Drug Resistant Active
MeSH Terms: interventions — OPC-67683; Linezolid; Levofloxacin; Pyrazinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- DAZZLE-24 wks (Experimental): Delamanid, Linezolid, Levofloxacin, Pyrazinamide (DAZZLE) treatment regimen- delamanid 100 mg PO BID, linezolid 600 mg PO QD, levofloxacin 1000 mg PO QD, and pyrazinamide 20-30 mg/Kg PO QD for 24 weeks, with linezolid dose reduction to 300 mg daily after 16 weeks (these doses are the usual doses for treatment of TB for all 4 study agents).
  Interventions: Drug: Delamanid; Drug: Linezolid; Drug: Levofloxacin; Drug: Pyrazinamide
- DAZZLE-32 wks (Experimental): Delamanid, Linezolid, Levofloxacin, Pyrazinamide (DAZZLE) delamanid 100 mg PO BID, linezolid 600 mg PO QD, levofloxacin 1000 mg PO QD, and pyrazinamide 20-30 mg/Kg PO QD for 32 weeks, with linezolid dose reduction to 300 mg daily after 16 weeks (these doses are the usual doses for treatment of TB for all 4 study agents).
  Interventions: Drug: Delamanid; Drug: Linezolid; Drug: Levofloxacin; Drug: Pyrazinamide
- DAZZLE-40 wks (Experimental): Delamanid, Linezolid, Levofloxacin, Pyrazinamide (DAZZLE) treatment regimen: delamanid 100 mg PO BID, linezolid 600 mg PO QD, levofloxacin 1000 mg PO QD, and pyrazinamide 20-30 mg/Kg PO QD for 40 weeks, with linezolid dose reduction to 300 mg daily after 16 weeks (these doses are the usual doses for treatment of TB for all 4 study agents).
  Interventions: Drug: Delamanid; Drug: Linezolid; Drug: Levofloxacin; Drug: Pyrazinamide
- DAZZLE-48 wks (Experimental): Delamanid, Linezolid, Levofloxacin, Pyrazinamide (DAZZLE) treatment regimen- delamanid 100 mg PO BID, linezolid 600 mg PO QD, levofloxacin 1000 mg PO QD, and pyrazinamide 20-30 mg/Kg PO QD for 48 weeks, with linezolid dose reduction to 300 mg daily after 16 weeks (these doses are the usual doses for treatment of TB for all 4 study agents).
  Interventions: Drug: Delamanid; Drug: Linezolid; Drug: Levofloxacin; Drug: Pyrazinamide
- DAZZLE-56 wks (Experimental): Delamanid, Linezolid, Levofloxacin, Pyrazinamide (DAZZLE) treatment regimen- delamanid 100 mg PO BID, linezolid 600 mg PO QD, levofloxacin 1000 mg PO QD, and pyrazinamide 20-30 mg/Kg PO QD for 56 weeks, with linezolid dose reduction to 300 mg daily after 16 weeks (these doses are the usual doses for treatment of TB for all 4 study agents).
  Interventions: Drug: Delamanid; Drug: Linezolid; Drug: Levofloxacin; Drug: Pyrazinamide
- WHO MDR-TB regimen- 9 mos or 20-24 mos (Active Comparator): MDR-TB treatment with 9-month or 20-24 month WHO approved regimen. The WHO guidelines recommend the following 5-agent treatment regimen for MDR-TB: pyrazinamide; a fluoroquinolone; a parenteral agent (typically amikacin or kanamycin); ethionamide (or prothionamide); and either cycloserine or para-aminosalicylic acid, with preference for cycloserine.
  Interventions: Drug: WHO MDR-TB regimen

INTERVENTIONS:
Drug: Delamanid — Delamanid is a medication used to treat tuberculosis. Specifically it is used, along with other antituberculosis medications, for active multidrug-resistant tuberculosis. It is taken by mouth.
  Other Names: Deltyba
  Arms: DAZZLE-24 wks; DAZZLE-32 wks; DAZZLE-40 wks; DAZZLE-48 wks; DAZZLE-56 wks
Drug: Linezolid — Linezolid is an antibiotic used for the treatment of infections caused by Gram-positive bacteria that are resistant to other antibiotics.
  Other Names: Zyvox
  Arms: DAZZLE-24 wks; DAZZLE-32 wks; DAZZLE-40 wks; DAZZLE-48 wks; DAZZLE-56 wks
Drug: Levofloxacin — Levoflaxacin is an antibiotic used to treat a number of bacterial infections including acute bacterial sinusitis, pneumonia, urinary tract infections, chronic prostatitis, and some types of gastroenteritis. Along with other antibiotics it may be used to treat tuberculosis.
  Other Names: Levaquin
  Arms: DAZZLE-24 wks; DAZZLE-32 wks; DAZZLE-40 wks; DAZZLE-48 wks; DAZZLE-56 wks
Drug: Pyrazinamide — Pyrazinamide is a medication used in combination with other drugs such as isoniazid and rifampicin in the treatment of Mycobacterium tuberculosis.
  Other Names: Zinamide
  Arms: DAZZLE-24 wks; DAZZLE-32 wks; DAZZLE-40 wks; DAZZLE-48 wks; DAZZLE-56 wks
Drug: WHO MDR-TB regimen — The WHO guidelines recommend the following 5-agent treatment regimen for MDR-TB: pyrazinamide; a fluoroquinolone; a parenteral agent (typically amikacin or kanamycin); ethionamide (or prothionamide); and either cycloserine or para-aminosalicylic acid, with preference for cycloserine. Short (9 mos) or longer (20-24 mos) treatment schedules can be used.
  Other Names: 5-agent treatment regimen for MDR-TB
  Arms: WHO MDR-TB regimen- 9 mos or 20-24 mos

SUMMARY:
The proposed study will randomize adults (18 years of age or older) with pulmonary MDR-TB with sputum that contains M. tuberculosis that is isoniazid and rifampin resistant by MTBDRplus and fluoroquinolone susceptible by MTBDRsl HIV seropositive (with or without antiretroviral therapy) or negative (but not unknown) and Karnofsky score of >60 at sites in Moldova, Peru, and the Philippines.

Patients with MDR-TB will be randomized to oral regimen of delamanid (DLM), linezolid (LZD), levofloxacin (LFX) and pyrazinamide (PZA) for 24, 32, 40, 48 or 56 weeks or World Health Organization (WHO) standard of care MDR-TB regimen (9-month "modified Bangladesh" regimen or WHO standard MDR-TB regimen).

Primary Objective

1. Determine the shortest duration of the delamanid-containing oral regimen that is non-inferior to the blended WHO standard regimen.

Secondary Objective

1. Define the safety and tolerability of the oral delamanid, linezolid, levofloxacin and pyrazinamide regimen.
2. Determine if baseline PZA susceptibility is associated with shorter time to non-inferior treatment duration.
3. Identify the relationship between delamanid and linezolid serum drug levels and time to sputum culture conversion among patients on the delamanid-containing oral regimen.
4. Identify the relationship between delamanid and linezolid serum drug levels and occurrence of adverse events among patients on the delamanid-containing oral regimen.

DETAILED DESCRIPTION:
Multidrug-resistant tuberculosis (MDR-TB) is tuberculosis that is resistant to at least isoniazid and rifampicin, the two most important anti-TB drugs. WHO has estimated that over 480,000 new cases of MDR-TB occurred in 127 countries in 2014, causing 150,000 deaths; this represents a 70% increase in the number of cases since 2000. MDR-TB cure rates are substantially lower than the 85+% cure expected in drug-susceptible TB. The MDR-TB treatment regimen currently recommended by WHO includes at least 4 second-line drugs plus PZA for 18-24 months, including an injectable agent for the induction phase of 6-8 month. However, the average global success rate of such treatment among patients treated in TB programs is only 50%. More recently, an alternative treatment regimen, known as the "Bangladesh" regimen, has become available.This regimen uses 7 drugs given for 9 months but still includes an injectable agent, which is the cause of the most common and severe toxicities seen when treating MDR-TB. In selected patients this regimen has been able to achieve over 80% cures, but use has been restricted to geographic areas where previous use of second-line drugs is rare. Alternatives will be necessary for other settings and patients with prior second-line drug exposure.

Treatment-limiting side effects are common when using second-line drugs for long periods of time. Overall, 69-73% of patients with MDR-TB treated with the WHO standard regimen are reported to have experienced at least one side effect, and 29%-55% discontinued one or more study drugs because of inability to tolerate a drug. The Bangladesh regimen also has substantial toxicity, with 63% of participants experiencing adverse drug reactions in one report. Thus, while this regimen is shorter and slightly better tolerated than the WHO standard regimen, it still does not provide an easily tolerated alternative, largely because it contains an injectable agent.

The 20-24 month regimen currently in use exposes patients to drug toxicity over prolonged periods of time and demands substantial human resources. Patients receiving these regimens require two years of directly observed therapy with careful monitoring for drug toxicity. Reduction in the duration of treatment would free up program staff to treat additional MDR-TB patients. Development of a shorter treatment regimen will greatly enhance the ability of programs to keep up with the anticipated increase in patients needing treatment.

This application proposes a study to determine whether the 9-month oral regime that uses Delaminid, Linezolid, Levofloxacin and Pyrazinamide is as good as the current WHO standard of care regimen.

The study proposes to randomize approximately 300 adults in Peru, Moldova and Phillipines where MDR-TB is common.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age ≥18 years
2. Subject has pulmonary TB
3. Sputum Smear, culture or Xpert MTB/RIF assay positive, with Hain MTBDRplus showing Rifampin (RIF) resistance and Isoniazid (INH) resistance and Hain MTBDRsl showing Fluoroquinolone susceptibility.
4. Patients within two weeks (≤14 days) of starting second-line anti-TB drugs
5. HIV seropositive or seronegative but not unknown HIV serostatus. If the last documented negative HIV test was more than 3 months prior to randomization the current serostatus must be assessed.
6. Karnofsky score of > 60 (see Appendix B) at screening and randomization
7. Willingness by the patient to attend scheduled follow-up visits and undergo study assessments.
8. Women with child-bearing potential must agree to practice an adequate birth control or to abstain from heterosexual intercourse during study regimen.
9. Laboratory parameters (performed within 14 days prior to randomization):

   * Estimated Serum creatinine < 2.0
   * Hemoglobin concentration ≥ 7.0 g/dL
   * Platelet count of ≥ 80,000/mm3
   * Absolute neutrophil count (ANC) > 2000/ mm3
   * Negative pregnancy test (for women of childbearing potential) during randomization/baseline
   * CD4 count if HIV infected (within 6 months)
   * Serum ALT and total bilirubin <3 times upper limit of normal
   * Serum albumin > 2.8 g/dL
10. Able to provide informed consent

Exclusion Criteria:

1. Known quinolone-resistance
2. History of serotonin syndrome
3. History of symptomatic arrhythmia, or taking anti-arrhythmic agents
4. Previous treatment with delamanid or linezolid
5. Known allergy or intolerability to quinolone or pyrazinamide
6. Patients who are pregnant or who are unwilling to use proper contraceptives at childbearing age
7. Medical history of galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
8. The need for ongoing use of prohibited drugs while on study drugs (see section 5.6 below)
9. History of optic neuropathy or peripheral neuropathy
10. History of hypersensitivity reaction to the study drugs
11. Patient is eligible for delamanid or bedaquiline under national program criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Successful outcome at 18 months after randomization using culture results, follow up visits, | 18 months
  Successful outcome:if they have a -ve liq culture result 18 mos post rand not having been prev. classified as unsuccessful. If pt unable to produce sputum at 18 mos, the outcome will be classified as successful if they have a -ve culture at last visit at which they were able to produce sputum. Unsuccessful outcome: any of the foll occur, if patient 1)d/c from allocated study treatment & restarted on a diff MDR-TB regimen; 2)has surgery for MDR-TB; 3)treatment extended beyond the scheduled end of treatment for any reason other than making up of missed treatment; 4)restarted on MDR-TB treatment post the sched end of treatment; 5)Allocated treatment changed for any reason other than d/c of PZA when isolate is resistant to PZA; 6)death at any point up to 18 mos post-rand; 7)has a +ve sputum culture 8 wks before the sched completion; 8)has +ve sputum culture after culture conversion by dates specified in criterion number 7; 9)ltfu at any time post rand & before completion of the 18 mos f/u

SECONDARY OUTCOMES:
Secondary - Adverse Events | 18 months
  Adverse Events (AE) grade 3 and above, regardless of relatedness to drugs in the patient's MDR-TB treatment regimen

CONTACTS AND LOCATIONS:
Overall Officials: C. Robert Horsburgh, MD, Principal Investigator — Boston University

IPD SHARING:
Plan to Share IPD: Undecided